CLINICAL TRIAL: NCT06647459
Title: Defining the Risk of Ventricular Tachycardia in Genetic Forms of Early-onset Atrial
Brief Title: Defining the Risk of Ventricular Tachycardia in Genetic Forms of Early-onset Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, M. Benjamin Shoemaker, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 231260
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ventricular Tachycardia; Atrial Fibrillation
Keywords: catheter ablation; genomics
MeSH Terms: conditions — Tachycardia, Ventricular; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pathogenic variant in TTN: 50 patients with a pathogenic variant in TTN
  Interventions: Diagnostic Test: EP Study
- Pathogenic variant in other cardiomyopathy genes: 50 patients with a pathogenic variant in other cardiomyopathy genes
  Interventions: Diagnostic Test: EP Study
- Genotype-negative controls: 100 genotype-negative controls
  Interventions: Diagnostic Test: EP Study

INTERVENTIONS:
Diagnostic Test: EP Study — To use programmed ventricular stimulation at the time of AF ablation to define the prevalence and mechanism of inducible ventricular tachycardia (VT); pace-mapping to define the site of origin of ventricular arrhythmias; and voltage mapping to define low voltage scar substrate in the basal LV in patients with pathogenic TTN variants compared to genotype-negative controls.
  Other Names: Mapping

SUMMARY:
To use programmed ventricular stimulation at the time of AF ablation to define the prevalence and mechanism of inducible ventricular tachycardia (VT); pace-mapping to define the site of origin of ventricular arrhythmias; and voltage mapping to define low voltage scar substrate in the basal LV in patients with pathogenic TTN variants compared to genotype-negative controls.

DETAILED DESCRIPTION:
Participants will undergo AF ablation according to standard, contemporary techniques. The procedure will be performed under general anesthesia. As part of routine standard of care in patients with early-onset AF or patients who have PVCs, we will also test for inducibility of VT using a standardized pacing protocol. The research protocol will include LV mapping and identification of low voltage substrate using electroanatomical mapping as described below.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and older
2. Diagnosed with AF before age 60
3. Scheduled for catheter-based AF ablation (de-novo or repeat)
4. Able to provide written, informed consent
5. P/LP variant in TTN or other CM gene (cases) or identified as a genotype-negative control.

Exclusion Criteria:

1. Diagnosed with a genetic CM or arrhythmia syndrome prior to AF
2. VUS in 'possibly pathogenic' subgroup (control group only)
3. Pacemaker or ICD
4. Previous PVC or VT ablation
5. LVEF <20%
6. Prosthetic mitral or aortic valve
7. Contraindication to heparin
8. Prior myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with early-onset AF are referred to our Vanderbilt AF Precision Medicine Clinic and undergo clinical genetic testing with a CM/arrhythmia panel and a comprehensive clinical evaluation including a cardiac MRI. 50% of patients are referred to undergo AF ablation to treat symptomatic AF. For all eligible patients, the study will be described either in person, or be contacted via phone with an approved phone script. If interested, participants sign the written informed consent (paper option or e-consent option).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
VT Inducibility | At the time of procedure
  The primary endpoint is induction of sustained VT that is determined to be reentrant or likely-reentrant. Sustained VT will be defined as VT lasting 30 seconds or requiring termination with burst pacing or cardioversion due to hemodynamic instability.
Presence of ventricular arrhythmias per specific site | At the time of procedure
  The primary endpoint is the occurrence (yes/no) of ventricular arrhythmias (PVCs, NSVT, sustained VT) that are mapped to the basal LV as defined above.
Low voltage substrate | At the time of procedure
  The primary endpoint is the presence of low voltage (yes/no) in the basal LV.

SECONDARY OUTCOMES:
Site of origin for ventricular arrhythmias | At the time of procedure
  Secondary analyses will explore the rate of ventricular arrhythmias in other segments of the LV and RV and will compare the site of origin for ventricular arrhythmias in the group of participants with pathogenic variants in other CM genes.
Evaluation of electrogram potentials | At the time of procedure
  Secondary analyses will explore multicomponent electrograms and fractionated potentials that can be created by scar.
Presence of low voltage | At the time of procedure
  Other secondary analyses will compare the presence of low voltage and the other secondary endpoints in the group of participants with pathogenic variants in other CM genes.

CONTACTS AND LOCATIONS:
Overall Officials: Moore B Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT06647459/ICF_001.pdf